CLINICAL TRIAL: NCT00015652
Title: A Pilot Study of Low Dose Interleukin-2 (IL-2) With the Addition of Pegylated Interferon (PEG-IFN Alfa-2b) and Ribavirin (RBV) for the Treatment of Hepatitis C Infection in Subjects With HIV Coinfection
Brief Title: Interleukin-2 (IL-2), Pegylated Interferon (PEG-IFN Alfa-2b), and Ribavirin (RBV) Treatment in Patients With Hepatitis C and HIV Coinfection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A5088; AACTG A5088; 10676 (Registry Identifier: DAIDS ES Registry Number); ACTG A5088
Record Dates: First submitted 2001-04-26; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Ribavirin; Polyethylene Glycols; Interferon Alfa-2b; Dose-Response Relationship, Drug; Drug Therapy, Combination; Antiviral Agents; Hepatitis C; Aldesleukin; Peginterferon
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Ribavirin; aldesleukin; peginterferon alfa-2b

INTERVENTIONS:
Drug: Ribavirin
Drug: Aldesleukin
Drug: Peginterferon alfa-2b

SUMMARY:
This study will test the safety and effectiveness of a new treatment for hepatitis C (HCV) in patients who also have HIV.

The usual treatment for HCV in people who are not HIV-infected is interferon-alfa (IFN) with ribavirin (RBV), an approved treatment by the Food and Drug Administration (FDA). This study will use a new, longer acting form of IFN called PEG-IFN alfa-2b. PEG-IFN alfa-2b is approved by the FDA for use in treating HCV but has not yet been approved for use with RBV. This study also will use IL-2, which is a substance that the body naturally produces. People with HIV infection usually do not make enough IL-2. IL-2 is being tested in this study to see if it will "boost" the immune system's response to HCV. The FDA has approved IL-2 for the treatment of some cancers.

DETAILED DESCRIPTION:
HCV infection is an increasingly important clinical problem in patients infected with HIV. In HIV-uninfected patients with acute HCV infection, the presence of vigorous T-cell proliferative responses to HCV proteins is associated with normalization of serum transaminase levels and viral clearance. Furthermore, early results suggest IL-2 may improve transaminase levels in HCV/HIV patients. These observations provide the rationale for an immune-based therapeutic approach to HCV/HIV coinfection. This study explores the use of initial immunostimulatory therapy with IL-2 followed by the addition of antiviral therapy with PEG-IFN alfa-2b and RBV, as a possible synergistic approach to treatment.

Patients receive IL-2 for 12 weeks followed by the addition of PEG-IFN alfa-2b and RBV at the Week 12 visit. Patients remain on IL-2, PEG-IFN alfa-2b, and RBV for an additional 48 weeks. At Week 60, all study treatment is permanently discontinued and patients continue to be evaluated through Week 84. Toxicity or intolerance is evaluated. Data is collected on biochemical and virologic responses.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are between 18 and 65 years of age.
* Are infected with HIV.
* Have been on the same anti-HIV drugs and doses, if on any, for 8 weeks or longer and intend to stay on these drugs the first 24 weeks of the study. If patients have not been on anti-HIV drugs, they should not start them during the first 24 weeks of the study.
* Have a CD4 count of 300 cells/mm3 or more within 30 days before study entry.
* Have an HIV viral load of less than 5,000 copies/ml within 30 days before study entry.
* Have a detectable HCV viral load within 30 days before study entry.
* Have a chronic HCV infection at least 6 months before study entry.
* Can document chronic hepatitis within 24 months before study entry.
* Agree not to become pregnant (females) or make someone pregnant (males), or donate sperm, or participate in any other fertilization procedures while on the study drugs and for 6 months afterwards. Agree to use reliable forms of birth control during the same time period.
* Have a negative pregnancy test within 30 days of study entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have IgM antibody to hepatitis A within 30 days before study entry.
* Are coinfected with HBV within 30 days before study entry.
* Have had a liver biopsy showing liver disease (unless due to HCV) within 2 years before study entry.
* Have disease associated with the immune system such as Crohn's disease, ulcerative colitis, active rheumatoid arthritis, lupus, idiopathic thrombocytopenic purpura, autoimmune hemolytic anemia, cryoglobulinemia with clinical manifestations including leukocytoclastic vasculitis, scleroderma, and severe psoriasis.
* Have severe cirrhosis of the liver.
* Have significant heart problems.
* Have a thyroid problem which has not been treated.
* Have a history of severe mental problems.
* Have taken the following within 6 weeks before study entry: rifampin, rifabutin, pyrazinamide, isoniazid, G-CSF (filgrastim), GM-CSF (sargramostim), or ganciclovir.
* Have taken any of the following within 6 months before study entry: interleukins, interferons, therapeutic HIV vaccine, thalidomide, pentoxifylline, dinitrochlorobenzene (DNCB), thymosin alpha, thymopentin inosiplex, polyribonucleoside, ditiocarb sodium, hydroxyurea, systemic corticosteroids, azathioprine, 6-mercaptopurine, cyclosporin A, or any investigational drug.
* Have taken interferon or ribavirin any time before study entry.
* Have a disease affecting the red blood cells.
* Have retinopathy (disease of the eye).
* Have a chronic liver disease other than HCV.
* Are pregnant or breast-feeding.
* Are allergic to IL-2, PEG-IFN alfa-2b, or RBV or other components of the study products.
* Are presently using illegal drugs.
* Have had more than 1 alcoholic drink per day during the previous 30 days before study entry, or more than 4 drinks per day during the previous 6 months.
* Have been treated for a serious infection or other serious medical illness within 14 days before study entry.
* Have uncontrolled seizures.
* Have serious breathing and lung problems.
* Have had a major organ transplantation.
* Have history of a severe medical problem that would make the patient unsuitable for the study.
* Have had treatment for cancer or treatment affecting the immune system within 24 weeks before study entry or expect to need such treatment at any time during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Glesby, Study Chair
Locations (8):
- United States (8):
  - UCLA CARE Center CRS, Los Angeles, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas